CLINICAL TRIAL: NCT05575297
Title: A Drug-drug Interaction Study to Evaluate the Effect of Rifampicin and Febuxostat on the Pharmacokinetics of Methotrexate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MRFI
Record Dates: First submitted 2022-10-04; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Methotrexate; Febuxostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methotrexate (Experimental)
  Interventions: Drug: Methotrexate Sodium
- Methotrexate + Rifampicin (Experimental): Methotrexate + Rifampicin
  Interventions: Drug: Methotrexate Sodium; Drug: Rifampicin Sodium
- Methotrexate + Febuxostat (Experimental): Methotrexate + Febuxostat
  Interventions: Drug: Methotrexate Sodium; Drug: Febuxostat Tablets
- Methotrexate + Rifampicin + Febuxostat (Experimental): Methotrexate + Rifampicin + Febuxostat
  Interventions: Drug: Methotrexate Sodium; Drug: Rifampicin Sodium; Drug: Febuxostat Tablets

INTERVENTIONS:
Drug: Methotrexate Sodium — Methotrexate oral administration alone
Drug: Rifampicin Sodium — Co-administration of methotrexate and rifampicin
  Arms: Methotrexate + Rifampicin; Methotrexate + Rifampicin + Febuxostat
Drug: Febuxostat Tablets — Co-administration of methotrexate and febuxostat
  Arms: Methotrexate + Febuxostat; Methotrexate + Rifampicin + Febuxostat

SUMMARY:
To investigate the effect of rifampicin and febuxostat on pharmacokinetics of methotrexate in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 50, healthy male subjects (at screening)
* Body weight between 50.0 kg - 90.0 kg, BMI between 18.0 - 30.0 kg/m2
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress

Exclusion Criteria:

* Subject who has a past or present history of any diseases (eg. liver, kidney, neurology, immunology, pulmonary, endocrine, hematology, oncology, cardiology, mental disorder)
* Subject who had GI tract disease (Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery (appendectomy, hernioplasty are excluded)
* Serum AST(SGOT), ALT(SGPT), total bilirubin >1.5 times upper limit of normal range, MDRD eGFR < 60mL/min/1.73m2, WBC count < 3,500 /uL, SBP < 90 mmHg or > 150 mmHg, DBP < 50 mmHg or >100 mmHg
* Subject who had galactose intolerance, Lapplactase deficiency or glucose-galactose malabsorption
* Subject who had received drugs inhibiting or inducing metabolic enzymes/transporters such as barbiturates, statins, digoxin in 3 months
* Subject who had taken St.John's wort and food including grapefruit in 2 weeks
* Smoking in 3 months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 month or transfusion in 1 month currently

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Compare Cmax of methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2, 3, 4 Day 1)
  Compare the maximum concentration (Cmax), area under the plasma concentration-time curve to last measurable time point (AUClast) and area under the plasma concentration-time curve from 0 hours to infinite time (AUCinf) of methotrexate
Compare AUClast of methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2, 3, 4 Day 1)
  Compare the area under the plasma concentration-time curve to from 0 to last measurable time point (AUClast) of methotrexate
Compare AUCinf of methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2, 3, 4 Day 1)
  Compare area under the plasma concentration-time curve from 0 hours to infinite time (AUCinf) of methotrexate

SECONDARY OUTCOMES:
Compare Cmax of 7-hydroxy methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2, 3, 4 Day 1)
  Compare the maximum concentration (Cmax) of 7-hydroxy methotrexate
Compare AUClast of 7-hydroxy methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2, 3, 4 Day 1)
  Compare area under the plasma concentration-time curve to last measurable time point (AUClast) of 7-hydroxy methotrexate
Compare AUCinf of 7-hydroxy methotrexate | pre-dose (0h), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24 h post-dose (Period 1, 2, 3, 4 Day 1)
  Compare area under the plasma concentration-time curve from 0 hours to infinite time (AUCinf) of 7-hydroxy methotrexate

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided